CLINICAL TRIAL: NCT05449015
Title: Study on the Effect of Two Ways of Cycloplegia on Biological Parameters of Ciliary Muscle
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2022SQ006
Record Dates: First submitted 2022-06-28; First posted 2022-07-08 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Accomodation; Refractive Errors; Myopia; Cycloplegia
MeSH Terms: conditions — Refractive Errors; Myopia | interventions — Atropine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1% atropine (Experimental): 1% atropine eye drops, in the conjunctival sac, once a night, for 7 days
  Interventions: Drug: 1% atropine
- tropicamide (Placebo Comparator): tropicamide eye drops, in the conjunctival sac, once every 5 minutes, after 3 consecutive doses, close eyes for 20 minutes
  Interventions: Drug: 1% atropine

INTERVENTIONS:
Drug: 1% atropine — Daily application can be used for mydriasis and refraction examination Weekly long-term application can be used to control myopia

SUMMARY:
Atropine has a ciliary muscle-paralysing effect and causes hyperopic drift. Besides, atropine has been proven to slow the progression of myopia. Many studies have suggested that atropine can increase the thickness of the choroid. However, few studies have discussed changes in the ciliary muscle after treatment with atropine or other cycloplegic agents.

This study aimed to assess the difference in ciliary muscle morphology before and after two different cycloplegic agents and to analyze the correlation between the changes of ciliary muscle biological parameters and the changes of eye axis, spherical equivalent, lens diopter, choroidal thickness, etc. One hundred and forty-four children would be randomly assigned 1:1 to the 1% atropine group and the tropicamide group. This study might provide clinical evidence for the role of regulatory factors in the occurrence and development of myopia.

DETAILED DESCRIPTION:
The ciliary muscle exhibited an inward-forward contraction during accommodation, resulting in a significant thickening of the anterior area of the ciliary muscle. In addition to ultrasound biomicroscope (UBM), anterior segment optical coherence tomography (AS-OCT) is also commonly used to study morphological changes in the ciliary muscle. Studies using AS-OCT revealed that the posterior area of the ciliary muscle thinned during accommodation.

The morphology of the ciliary muscles differs in individuals with refractive errors. Many researchers found that the ciliary muscle became thicker with an increase of axial length (AL) Some studies suggested that myopia primarily affected the posterior area of the ciliary muscle.

Atropine has a ciliary muscle-paralysing effect and causes hyperopic drift. Besides, atropine has been proven to slow the progression of myopia. Many studies have suggested that atropine can increase the thickness of the choroid. However, few studies have discussed changes in the ciliary muscle after treatment with atropine or other cycloplegic agents.

This study aimed to assess the difference in ciliary muscle morphology before and after two different cycloplegic agents and to analyze the correlation between the changes of ciliary muscle biological parameters and the changes of eye axis, spherical equivalent, lens diopter, choroidal thickness, etc. One hundred and forty-four children would be randomly assigned 1:1 to the 1% atropine group and the tropicamide group. This study might provide clinical evidence for the role of regulatory factors in the occurrence and development of myopia.

ELIGIBILITY:
Inclusion Criteria:

* ①Age 3 to 12 years old;

  * Astigmatism <2.00D, binocular anisometropia <3.00D, and the best corrected distance visual acuity is at least 0.8, near vision at least 0.8;

    * A clear anterior segment image can be obtained through anterior segment OCT;

      * Have normal thinking and language communication skills, and can actively cooperate with the inspection process; ⑤ No contraindications to atropine treatment such as acute eye inflammation, dry eye, keratoconus, diabetes, etc.; ⑥Written informed consent of the guardian and the child himself

Exclusion Criteria:

* ① Combined with neurological diseases and have allergies or contraindications to cycloplegic drugs or other drugs;

  * Intraocular pressure ≥21mmHg; history of photosensitivity, glaucoma, blue eye syndrome, ocular hypertension, and retinal macular lesions or damage;

    * Patients with chronic eye diseases such as ocular trauma and allergic conjunctivitis;

      * Those who wear contact lenses and those who use myopia control-related drugs within 1 month; ⑤ Patients with previous varus trichiasis, severe horn, conjunctiva infection and other eye diseases;

        * Insufficient image quality, such as inconsistent field of view, poor image exposure, inaccurate image focus, stains, shadows or crescent shadows, etc.;

          * There are systemic diseases; ⑧ Epilepsy, mental disorders unable to communicate normally; ⑨ Other circumstances judged by the investigator to be unsuitable to participate in the research

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
ciliary thickness parameters | before intervention
  ciliary thickness parameters, microns(um), photographed by ASOCT and measured by semiautomatic software
ciliary thickness parameters | immediately after the last intervention
  ciliary thickness parameters, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | before intervention
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software
the distance between ciliary muscle apex and scleral spur | immediately after the last intervention
  ciliary muscle thickness, microns(um), photographed by ASOCT and measured by semiautomatic software

SECONDARY OUTCOMES:
spherical equivalent | before intervention
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
spherical equivalent | immediately after the last intervention
  spherical equivalent(SE)，Diopter(D), measured by subjective optometry
axial length | before intervention
  axial length(AL), millimeter(mm), measured by IOL master
axial length | immediately after the last intervention
  axial length(AL), millimeter(mm), measured by IOL master

OTHER OUTCOMES:
choroidal thickness | before intervention
  choroidal thickness, microns(um), measured by SSOCT
choroidal thickness | immediately after the last intervention
  choroidal thickness, microns(um), measured by SSOCT
lens thickness | before intervention
  lens thickness(LT), millimeter(mm), measured by IOL master
lens thickness | immediately after the last intervention
  lens thickness(LT), millimeter(mm), measured by IOL master
lens power | before intervention
  lens power(LP), diopter(D), calculated by Bennett formula
lens power | immediately after the last intervention
  lens power(LP), diopter(D), calculated by Bennett formula
corneal parameters | before intervention
  central corneal thickness(CTC), micron(um), measured by IOL master
corneal parameters | immediately after the last intervention
  central corneal thickness(CTC), micron(um), measured by IOL master
retinal thickness | before intervention
  retina thickness, microns(um), measured by SSOCT
retinal thickness | immediately after the last intervention
  retina thickness, microns(um), measured by SSOCT

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Zou, M.D., Study Director — Shanghai Eye Diseases Prevention Treatment Center
Locations (1):
- Shanghai Eye Diseases Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT05449015/Prot_000.pdf